CLINICAL TRIAL: NCT05854251
Title: Hyperinsulinemia in Prediabetes Mediated by Interleukin-1β- The Hyper-PreDIL-Study
Brief Title: Hyperinsulinemia in Prediabetes Mediated by Interleukin-1β
Acronym: Hyper-PreDIL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-00497; kt23Donath2
Record Dates: First submitted 2023-05-02; First posted 2023-05-11 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Hyperinsulinemia; PreDiabetes
Keywords: anakinra (Kineret®)
MeSH Terms: conditions — Hyperinsulinism; Prediabetic State | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Intervention Model Description: Placebo controlled, double-blind, randomized, cross-over proof-of-concept study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Intervention (Experimental): Patients receive investigational product
  Interventions: Drug: Anakinra
- Control Intervention (Placebo Comparator): Patients receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anakinra — Subjects receive an s.c. injection of 100 mg Anakinra on the evening before and on the respective study day 60 minutes before ingestion of the mixed-meal
  Arms: Experimental Intervention
Drug: Placebo — 0.67 ml of s.c. injection of saline will be taken on the evening before and on the respective study day 60 minutes before ingestion of the mixed-meal
  Arms: Control Intervention

SUMMARY:
The goal of this clinical study is to test whether postprandial insulin secretion in subjects with prediabetes is mediated by Interleukin-1β and may be influenced by administration of the medicinal product anakinra (Kineret®).

The main question it aims to answer is whether there is a difference in insulin secretion following a standardized mixed-meal test under anakinra compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with prediabetes defined by HbA1c 5.7-6.4 % or fasting plasma glucose 6.1-6.9 mmol/l or plasma glucose 2 h following 75g glucose ingestion of 7.8-11.0 mmol/l.
* BMI ≥ 28 kg/m2
* Age ≥ 18 years
* C-reactive protein ≥ 2 mg/dl
* For subjects with reproductive potential, willingness to use contraceptive measures adequate to prevent the subject from becoming pregnant during the study

Exclusion Criteria:

* Upper gastrointestinal surgery
* Diagnosis of any type of diabetes mellitus
* Signs of current infection
* Use of any glucose lowering medication within the last three months
* Use of investigational drug up to one week prior to start of treatment phase.
* Anti-inflammatory medication, including systemic glucocorticoid therapy.
* Neutropenia (leukocyte count < 1.5 × 109/L or absolute neutrophil count (ANC) < 0.5 × 109/L)
* Anemia (hemoglobin < 11 g/dL for males, < 10 g/dL for females)
* Clinically significant kidney or liver disease (creatinine > 1.5 mg/dL, aspartate aminotransferase (AST)/ alanine aminotransferase (ALT) > 2 × ULN, alkaline phosphatase > 2 × ULN, or total bilirubin [tBili] > 1.5 × ULN)
* Uncontrolled disease
* Currently pregnant or breastfeeding
* No subjects meeting the criteria for vulnerability. Participation in another study with investigational drug within the 30 days preceding and during the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Change in insulin concentration following a standardized mixed-meal test | two time assessment at baseline and after 1-2 weeks
  Changes in insulin concentration (mmol/l) under anakinra compared to placebo. Blood will be analysed 90 and 0 min before and 30 min, 1 hr, 1.5 hrs, 2 hrs, 2.5 hrs, 3 hrs after the mixed meal.
Change in glucose concentration following a standardized mixed-meal test | two time assessment at baseline and after 1-2 weeks
  Changes in glucose concentration (mmol/l) under anakinra compared to placebo. Blood will be analysed 90 and 0 min before and 30 min, 1 hr, 1.5 hrs, 2 hrs, 2.5 hrs, 3 hrs after the mixed meal.
Change in c-peptide concentration following a standardized mixed-meal test | two time assessment at baseline and after 1-2 weeks
  Changes in c-peptide concentration (nmol/l) under anakinra compared to placebo. Blood will be analysed 90 and 0 min before and 30 min, 1 hr, 1.5 hrs, 2 hrs, 2.5 hrs, 3 hrs after the mixed meal.
Change in insulinogenic index (IGI) concentration following a standardized mixed-meal test | two time assessment at baseline and after 1-2 weeks
  Changes in insulinogenic index (IGI) (I30 - I0)/(G30 - G0) under anakinra compared to placebo.
  Blood will be analysed 90 and 0 min before and 30 min, 1 hr, 1.5 hrs, 2 hrs, 2.5 hrs, 3 hrs after the mixed meal.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Donath, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland